CLINICAL TRIAL: NCT02951481
Title: Antimicrobial Stewardship Program Based on the Detection and Monitoring of Patients With Clostridium Difficile Infection (PACTA-ICD)
Brief Title: Antimicrobial Stewardship Program for Clostridium Difficile Infection.
Acronym: PACTA-ICD
Status: Completed | Type: Observational
Sponsor: José María Aguado García, MD, PhD (Other)
Collaborators: Hospital Universitario 12 de Octubre (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, José María Aguado García, MD, PhD, José María Aguado García, MD, PhD, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Other Study IDs: JMA-MET-2016-01
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Results first posted 2020-10-29 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Clostridium Difficile; Enterocolitis, Pseudomembranous
Keywords: Clostridium difficile.; Antimicrobial Stewardship.; Enterocolitis, Pseudomembranous
MeSH Terms: conditions — Enterocolitis, Pseudomembranous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — As patients with CDI are going to be prospectively followed, apart from the routine hematology and biochemistry analysis, serum immunoglobulin levels, serum complement levels (C3 and C4) and peripheral blood lymphocyte subpopulations will be measured at the end of CDI treatment.
  The levels of these immunological parameters will be tested as markers for relapse by retrospectively comparing them between patients with and without recurrence.
  A stool sample will be collected at the end of treatment to evaluate predictors of bad outcome or recurrence: Inflammatory markers (lactoferrin, calprotectin) We will retrospectively compare these parameters between patients with and without recurrence.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Systematic evaluation by an ID expert.: Patients diagnosed with CDI during 2017 in the University Hospital 12 de Octubre will be systematically evaluated by an Infectious Disease expert to ensure compliance with clinical practice guidelines about specific treatment for CDI, depending on the severity of the episode and the existence of previous episodes. This group of patients will also receive a close follow up during the period of greatest risk of relapse (8 weeks after completion of antibiotic treatment for CDI) in order to reduce as far as possible, the number of relapses.
  Interventions: Behavioral: Systematic evaluation by an ID expert.
- Retrospective historic cohort.: Patients diagnosed with CDI during 2015 in the University Hospital 12 de Octubre in which a systematic intervention was not done.

INTERVENTIONS:
Behavioral: Systematic evaluation by an ID expert. — Specific "bundle" of measures:
  1. Systematic evaluation of all patients diagnosed with CDI by an Infectious Disease expert To ensure compliance with clinical practice guidelines about specific treatment for CDI, depending on the severity of the episode and the existence of previous episodes and to optimize concomitant antibiotic therapy ("antimicrobial stewardship").
  2. To ensure appropriate monitoring during the period of greatest risk of relapse in order to reduce as far as possible, the number of relapses. Personalized assistance by telephone or by email for early consultation in case of recurrence of symptoms or need for a new antibiotic course.
  Groups: Systematic evaluation by an ID expert.

SUMMARY:
The purpose of this study is to determine whether a bundle of measures specifically designed for patients with ICD and applied by and Infectious Diseases expert during a year period (2017) will improve the prognosis and reduce the rate of recurrence, compared with the baseline phase (2015) in which no intervention was made.

DETAILED DESCRIPTION:
Patients with CDI benefit from the assessment and monitoring by an Infectious Diseases (ID) expert. Early intervention in patients diagnosed with a first episode of CDI would reduce the unnecessary use of antibiotics, improve prognosis by ensuring compliance with the clinical practice guidelines and reduce the number of recurrences.

Primary objective:

• To improve the prognosis of patients with CDI hospitalized during the period of intervention:

* Increasing the compliance with clinical practice guidelines about specific treatment for CDI (for the episode that generated the intervention), depending on the severity of the episode and the existence of previous episodes
* Reducing the recurrence rate by means of a close follow-up during the period of higher risk, avoiding factors that are known to predispose to recurrence.

Secondary objectives:

* To discontinue or to reduce the spectrum of unnecessary antibiotic treatments in this population ("antimicrobial stewardship"), especially during the episode of CDI and during the following 8 weeks.
* To discontinue inappropriate treatment of asymptomatic patients colonized by Clostridium difficile.
* To identify clinical and biological markers that could be used as predictors of recurrence.
* To identify patients with a high number of recurrences, that could benefit from novel or experimental treatments.

MATERIAL AND METHODS:

The first 100 patients fulfilling the inclusion criteria will be included in the study.

They will be retrospectively compared with the first 100 patients diagnosed with CDI during de previous year (2015) in which there was not a systematical intervention by a member of the Infectious Diseases Unit.

Specific "bundle" of measures for patients with ICD:

This measures are based in well-known and evidence-based elements that reduce the incidence and limit the spreading of Clostridium difficile:

* Systematic evaluation of all patients diagnosed with CDI by an Infectious Disease expert with the implementation of the following interventions:

  * To ensure compliance with clinical practice guidelines about specific treatment for CDI, depending on the severity of the episode and the existence of previous episodes, thus improving the prognosis of these patients and avoiding side effects.
  * To optimize concomitant antibiotic therapy (antimicrobial stewardship) through the following interventions: remove unnecessary treatments, shorten antibiotic courses as far as possible and avoid, if possible, broad-spectrum or high risk for developing CDI antibiotics.
  * To reduce indiscriminate use of proton-pump inhibitors or H2 receptor antagonists.
  * To provide clear instructions to patients and their families about the measures that should be implemented at home after discharge. To answer their questions and calm their fears about the CDI and need for isolation.
* To ensure appropriate monitoring during the period of greatest risk of relapse (8 weeks after completion of antibiotic treatment for CDI) in order to reduce as far as possible, the number of relapses by the following interventions:

  * Personalized assistance by telephone or by email for early consultation in case of recurrence of symptoms, in order to make:

    * Early diagnostic of relapses.
    * Appropriate treatment of subsequent episodes.
    * Detection of patients who could benefit from fecal microbiota transplantation.
    * Personalized assistance by telephone or by email for consultation in case of necessity of a new antibiotic course in order to:
    * Avoid unnecessary antimicrobial treatments.
    * Choose the antibiotic class with less risk of selecting C. difficile.
    * Evaluate preventive measures in an attempt to prevent the development of CDI.

Study timetable

* Patients will be evaluated by a member of the research team at CDI diagnosis. Specific treatment will be revised by the investigator with patient's physician in order to adapt it to the clinical guidelines, depending on the severity of the episode and the existence of previous episodes. Concomitant antibiotic treatments will be dropped or adjusted if possible. It is important to clarify that the study investigator will always make a suggestion according to the current evidence, but the final decision about treatment will be always made by patient's physician in charge.
* At the end of CDI treatment patient will be evaluated again by phone or at the outpatient's clinic in order to ensure resolution of symptoms and detect possible adverse events.

  o In this moment, a blood test will be performed in all study patients including: Full blood count, basic biochemistry analysis, Iron metabolism parameters: total iron-binding capacity, total serum iron, ferritin and transferrin. Nutritional parameters. Inflammatory markers: C-reactive protein and erythrocyte sedimentation rate. Serum immunoglobulin levels, serum complement levels (C3 and C4) and peripheral blood lymphocyte subpopulations.
* Beyond that point, there will be a personalized assistance by telephone or by email once a week until 8 weeks after the end of treatment.
* In case of recurrence of symptoms, need for admission or a new antimicrobial treatment, patient will be seen at the outpatient's clinic and will receive and individualized advice in order to achieve an early diagnose of relapse and to reduce the risk of recurrence.

Definitions:

Diarrhoea: Loose stools, i.e. taking the shape of the receptacle or corresponding to Bristol stool chart types 5-7, plus a stool frequency of three stools in 24 or fewer consecutive hours or more frequently than is normal for the individual.

An episode of CDI is defined as: A clinical picture compatible with CDI and microbiological evidence of free toxins and the presence of C. difficile in stool without reasonable evidence of another cause of diarrhoea or Pseudomembranous colitis as diagnosed during endoscopy, after colectomy or on autopsy.

Mild or moderate CDI: Diarrhoea without systemic symptoms, leukocytosis with a white blood cell count lower than15,000 cells/mL and a serum creatinine level less than 1.5 times the premorbid level.

Severe CDI: systemic symptoms of infection and/or leukocytosis with a white blood cell count of 15,000 cells/mL or higher or a serum creatinine level greater than or equal to 1.5 times the premorbid level.

Severe Complicated CDI: was defined by the presence of severe disease accompanied by life-threatening conditions such as ileus, toxic megacolon, refractory hypotension and/or multi-organ failure attributable to CDI.

Ileus: Signs of severely disturbed bowel function such as vomiting and absence of stool with radiological signs of bowel distension.

Toxic megacolon: Radiological signs of distension of the colon (>6 cm in transverse width of colon) and signs of a severe systemic inflammatory response (nausea, vomiting, dehydration, lethargy or tachycardia addition to fever and abdominal pain).

Leukocyte count to consider severity of the CDI: Any white blood cell count (WBC) measured between two days before and two days following the date of the stool sample. If a patient had WBC measured on the date of the stool sample then this was selected. If they did not have WBC measured on the date of the stool sample but had WBC measured between one day before and one day following their stool sample, then this was selected. If they did not have WBC measured between one day before and one day following their stool sample but had WBC measured between two days before and two days following their stool sample, then this was selected. If they did not have WBC measured on the date of the stool sample but had WBC measured both one day before and one day following the date of stool sample, or had WBC measured both two days before and two days after the stool sample but not between these measurements, then the highest of the two measurements was selected.

Definition of treatment response: Treatment response is present when either stool frequency decreases or stool consistency improves and parameters of disease severity (clinical, laboratory, radiological) improve and no new signs of severe disease develop.

Definition of recurrent CDI: Recurrence is present when CDI re-occurs within 8 weeks of successfully completing treatment for CDI.

Duration of diarrhea: was the sum of days from day 1 to the last day with diarrhea, followed by 2 or more days without diarrhea.

Antibiotics of high, medium and low risk for CDI: according to the table proposed by Aldeyab et al (S3. J Antimicrob Chemother 2012; 67: 2988-2996).

Data collection and analysis Patients in the pre-intervention period will be retrospectively identified from data microbiology (all isolates of Clostridium difficile of 2015 will be revised). Patients in the intervention period will be identified and prospectively followed by a member of the research team.

The variables will be collected in a coded database for further analysis.

Sample size calculation We present an exploratory study which aim is to evaluate the impact of an intervention, consisting on a bundle of measures for patients diagnosed with a first episode of CDI. The bundle includes antimicrobial stewardship, close follow-up, optimization of specific treatment for CDI and potential search for clinical and biological markers of recurrence.

The required sample size was estimated under the hypothesis that the application of a strategy based on a bundle to improve the management of CDI, would decrease the risk of recurrence as compared to the usual care performed in the retrospective period.

A recent review that evaluated the frequency of treatment failure and recurrence of CDI showed a recurrence rate after metronidazole treatment of 27.6% in studies performed in Europe during the previous 10 years.

Based in the previous literature, we expected a cumulative incidence of recurrence in the control group of 27.6%. The study would require a sample size of 99 for each group (i.e. a total sample size of 198, assuming equal group sizes), to achieve a power of 80% for detecting a reduction in proportions of 0.15 between the two groups (reference group - intervention) at a two sided p-value of 0.05.

Statistical Plans In 2014, in our institution 188 new cases of CDI were diagnosed. We assume that approximately 30% were recurrences of previous cases, so we extrapolate than 1 year will be enough to achieve the estimated sample size of 100 patients for the prospective period.

The data of qualitative variables will be expressed as absolute values and relative frequencies. The data of quantitative variables will be shown as mean ± standard deviation should be demonstrated normal distribution or median with interquartile range otherwise. Categorical variables will be compared using X ^ 2 or Fisher's exact test. Continuous variables will be compared using the Student's t-test or the Mann-Whitney U test. Statistical analysis will be conducted using SPSS version 15.0 (SPSS Inc, Chicago, Illinois, USA).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with CDI in the University Hospital "12 de Octubre", Madrid, Spain, requiring hospitalization or emergency room admission longer than 48 hours, from the beginning of the study on (estimated start date: January 2017).
* Patient or his/her representative sign the inform consent

Exclusion Criteria:

* Patients younger than 18 years of age.
* Patients with the diagnosis of inflammatory bowel disease.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with CDI during 2015 in the University Hospital 12 de Octubre (retrospective historic cohort) or adult patients diagnosed with CDI during 2017 in the University Hospital 12 de Octubre (prospective cohort in which intervention was made).
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose María Aguado, MD. PhD, Principal Investigator — University Hospital 12 de Octubre. Head of Infectious Disease Unit.
Locations (1):
- Unidad de Enfermedades Infecciosas. Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Debast SB, Bauer MP, Kuijper EJ; European Society of Clinical Microbiology and Infectious Diseases. European Society of Clinical Microbiology and Infectious Diseases: update of the treatment guidance document for Clostridium difficile infection. Clin Microbiol Infect. 2014 Mar;20 Suppl 2:1-26. doi: 10.1111/1469-0691.12418. PMID 24118601
- [Background] Srigley JA, Brooks A, Sung M, Yamamura D, Haider S, Mertz D. Inappropriate use of antibiotics and Clostridium difficile infection. Am J Infect Control. 2013 Nov;41(11):1116-8. doi: 10.1016/j.ajic.2013.04.017. Epub 2013 Aug 7. PMID 23932828
- [Background] Vonberg RP, Kuijper EJ, Wilcox MH, Barbut F, Tull P, Gastmeier P; European C difficile-Infection Control Group; European Centre for Disease Prevention and Control (ECDC); van den Broek PJ, Colville A, Coignard B, Daha T, Debast S, Duerden BI, van den Hof S, van der Kooi T, Maarleveld HJ, Nagy E, Notermans DW, O'Driscoll J, Patel B, Stone S, Wiuff C. Infection control measures to limit the spread of Clostridium difficile. Clin Microbiol Infect. 2008 May;14 Suppl 5:2-20. doi: 10.1111/j.1469-0691.2008.01992.x. PMID 18412710
- [Background] Aldeyab MA, Kearney MP, Scott MG, Aldiab MA, Alahmadi YM, Darwish Elhajji FW, Magee FA, McElnay JC. An evaluation of the impact of antibiotic stewardship on reducing the use of high-risk antibiotics and its effect on the incidence of Clostridium difficile infection in hospital settings. J Antimicrob Chemother. 2012 Dec;67(12):2988-96. doi: 10.1093/jac/dks330. Epub 2012 Aug 16. PMID 22899806
- [Background] Slayton RB, Scott RD, Baggs J, Lessa FC, McDonald LC, Jernigan JA. The cost-benefit of federal investment in preventing Clostridium difficile infections through the use of a multifaceted infection control and antimicrobial stewardship program. Infect Control Hosp Epidemiol. 2015 Jun;36(6):681-7. doi: 10.1017/ice.2015.43. Epub 2015 Mar 18. PMID 25783204

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Retrospective period recruitment: 2015 (12 months). Prospective period: from February 15, 2017 to December 15, 2017 (10 months)
Pre-assignment Details: The initial idea was to include overall a minimun 200 patients (100 per group). As 231 patients fulfilled the criteria to be included in the retrospective arm, we finally recruited 172 patients during the prospective period (with a systematical intervention). Due to the study design, all started patients completed the study. So, counting the two groups, 403 patients started and completed the study. Neither the retrospective arm nor the prospective one suffered losses.
Groups:
- Retrospective Historic Cohort: During 2015 (12 months), there were 231 patients with a first episode of CDI.
- Prospective Group: Patients diagnosed with a first episode of CDI in the University Hospital "12 de Octubre", Madrid, Spain, requiring hospitalization or emergency room admission longer than 48 hours, from the beginning of the study on (1-February-2017). From February 15, 2017 to December 15, 2017 (10 months) there were 172 patients diagnosed with with a first episode of CDI.
Period: Overall Study
Arm/Group | Retrospective Historic Cohort | Prospective Group
Started | 231 | 172
Completed | 231 | 172
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group (Prospective): Patients diagnosed with a first episode of CDI in the University Hospital "12 de Octubre", Madrid, Spain, requiring hospitalization or emergency room admission longer than 48 hours, from the beginning of the study on (1-February-2017). An intervention was made.
- Total: Total of all reporting groups
Arm/Group | Retrospective Historic Cohort. | Intervention Group (Prospective) | Total
Number analyzed (Participants) | 231 | 172 | 403
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.26 (19.36) | 64.73 (18.98) | 64.46 (19.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 96 | 218
  Male | 109 | 76 | 185
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Spain | 231 | 172 | 403
Previous Comorbidities [Count of Participants; unit: Participants]
  Diabetes mellitus | 37 | 38 | 75
  Solid organ transplantation | 21 | 32 | 53
  Chronic renal failure | 41 | 42 | 83
  Any immunocompromising condition | 70 | 48 | 118
  Inflammatory bowel disease | 17 | 9 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clostridium Difficile Infection Recurrence.
Description: Number of patients with a Clostridium difficile infection recurrence in each group within the following 8 weeks after the end of specific treatment for the initial Clostridium difficile infection episode.
Time Frame: Within 8 weeks after the end of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective Historic Cohort. | Intervention Group (Prospective)
Number analyzed (Participants) | 231 | 172
Participants | 34 | 21
Statistical Analysis 1: Comparison: Retrospective Historic Cohort. vs Intervention Group (Prospective); Test type: Superiority; p = 0.56, Chi-squared

2. Secondary Outcome: Number of Participants Experiencing More Than One Clostridium Difficile Infection Recurrence.
Description: Number of patients in each group who suffer from at least one recurrence within the following 8 weeks after the end of specific treatment for the first recurrence of Clostridium difficile infection.
Time Frame: 8 weeks after the end of specific treatment for the first recurrence of Clostridium difficile infection.
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective Historic Cohort. | Intervention Group (Prospective)
Number analyzed (Participants) | 231 | 172
Participants | 11 | 5
Statistical Analysis 1: Comparison: Retrospective Historic Cohort. vs Intervention Group (Prospective); Test type: Superiority; p = 0.55, Fisher Exact

3. Secondary Outcome: Number of Participants With The Right Choice Anti-Clostridium Difficile Infection Treatment (According to the Current Guidelines for Treatment of C. Difficile Infection).
Description: Our definition of right choice was judged according to the European Society of Clinical Microbiology and Infectious Diseases, 2013 and Clinical practice guidelines for Clostridium difficile infection in adults and children: 2017 update by the Infectious Diseases Society of America (IDSA) and Society for Healthcare Epidemiology of America (SHEA).
  * Right choice: According to the current guidelines, the medication is effective for the condition an also used at optimal doses and duration, without duplication or association with unnecessary drugs.
  * Inappropriate/suboptimal prescription: Overuse: inclusion of unnecessary medication for the condition, which may result in an increased risk of adverse reactions, drug-drug interactions and increased costs. Underuse: omission of a drug when there is a clear indication and no contraindications. The failure to prescribe essential medications may result in the worsening of the illness or therapeutic failure.
Time Frame: In the following 48 hours to the positive diagnostic result.
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective Historic Cohort. | Intervention Group (Prospective)
Number analyzed (Participants) | 231 | 172
Participants | 149 | 130
Statistical Analysis 1: Comparison: Retrospective Historic Cohort. vs Intervention Group (Prospective); Test type: Superiority; p = 0.023, Chi-squared

4. Secondary Outcome: Number of Participants With a Clostridium Difficile Infection That Received an Inappropriate Prescription by Overuse.
Description: Our definition of right choice of treatment was judged according to the European Society of Clinical Microbiology and Infectious Diseases, 2013 and Clinical practice guidelines for Clostridium difficile infection in adults and children: 2017 update by the Infectious Diseases Society of America (IDSA) and Society for Healthcare Epidemiology of America (SHEA).
  Inappropriate/suboptimal prescription: Overuse: inclusion of unnecessary medication for the condition, which may result in an increased risk of adverse reactions, drug-drug interactions and increased costs.
Time Frame: In the following 48 hours to the positive diagnostic result.
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective Historic Cohort. | Intervention Group (Prospective)
Number analyzed (Participants) | 231 | 172
Participants | 40 | 10
Statistical Analysis 1: Comparison: Retrospective Historic Cohort. vs Intervention Group (Prospective); Test type: Superiority; p < 0.001, Chi-squared

5. Secondary Outcome: Number of Participants With a Clostridium Difficile Infection That Received an Inappropriate Prescription by Underuse.
Description: Our definition of right choice was judged according to the European Society of Clinical Microbiology and Infectious Diseases, 2013 and Clinical practice guidelines for Clostridium difficile infection in adults and children: 2017 update by the Infectious Diseases Society of America (IDSA) and Society for Healthcare Epidemiology of America (SHEA).
  Inappropriate/suboptimal prescription: Underuse: omission of a drug when there is a clear indication and no contraindications. The failure to prescribe essential medications may result in the worsening of the illness or therapeutic failure.
Time Frame: In the following 48 hours to the positive diagnostic result.
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective Historic Cohort. | Intervention Group (Prospective)
Number analyzed (Participants) | 231 | 172
Participants | 15 | 10
Statistical Analysis 1: Comparison: Retrospective Historic Cohort. vs Intervention Group (Prospective); Test type: Superiority; p = 0.5, Chi-squared

6. Secondary Outcome: Number of Participants With Antimicrobial Adjustment.
Description: Percentage of patients with antibiotic treatments removed or adjusted as a result of the diagnosis of CDI.
Time Frame: In the following 2 weeks to the positive diagnostic result.
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective Historic Cohort. | Intervention Group (Prospective)
Number analyzed (Participants) | 231 | 172
Participants | 62 | 33
Statistical Analysis 1: Comparison: Retrospective Historic Cohort. vs Intervention Group (Prospective); Test type: Superiority; p = 0.07, Chi-squared

7. Secondary Outcome: All Cause Mortality
Description: Percentage of patients who die within 8 weeks of the Clostridium difficile infection diagnosis.
Time Frame: 8 weeks after the positive diagnostic result.
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective Historic Cohort. | Intervention Group (Prospective)
Number analyzed (Participants) | 231 | 172
Participants | 18 | 17
Statistical Analysis 1: Comparison: Retrospective Historic Cohort. vs Intervention Group (Prospective); Test type: Superiority; p = 0.47, Chi-squared

8. Secondary Outcome: Clostridium Difficile Infection Attributable Mortality Rate.
Description: Percentage of patients who die within 30 days of the Clostridium difficile infection diagnosis. CDI-attributable mortality denotes the judgment by investigators that the patient would not have died within 30 days with the absence of CDI. Medical data were retrospectively reviewed by two independent investigators with clinical experience in CDI. In case of discrepancy, a third expert was consulted.
Time Frame: 30 days after the positive diagnostic result.
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective Historic Cohort. | Intervention Group (Prospective)
Number analyzed (Participants) | 231 | 172
Participants | 11 | 4
Statistical Analysis 1: Comparison: Retrospective Historic Cohort. vs Intervention Group (Prospective); Test type: Superiority; p = 0.29, Fisher Exact

ADVERSE EVENTS:
Time Frame: 8 weeks after the positive diagnostic result
Arm/Group | Retrospective Historic Cohort. | Intervention Group (Prospective)
All-Cause Mortality (participants affected / at risk) | 18/231 | 17/170
Serious Adverse Events (participants affected / at risk) | 0/231 | 0/170
Other Adverse Events (participants affected / at risk) | 0/231 | 0/170

LIMITATIONS AND CAVEATS:
The main limitation could be that both populations (retrospective group and group of intervention) are not totally comparable and the change in recommendations over time between the 2 periods.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-02-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT02951481/Prot_SAP_000.pdf
  • Informed Consent Form (2016-02-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT02951481/ICF_001.pdf